CLINICAL TRIAL: NCT01070433
Title: A Phase II, Randomized, Controlled, Multi-Center Study of the Safety and Efficacy of Topically Applied MEBO Wound Ointment Compared to Standard of Care in Subjects With Diabetic Foot Ulcers
Brief Title: A Clinical Study of the Safety and Efficacy of MEBO Wound Ointment in Subjects With Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Skingenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEBO-DFU-PII-001 v. 4.0
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot Ulcers (DFUs)
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEBO Wound Ointment (MEBO) (Experimental): Topical application twice a day
  Interventions: Drug: MEBO Wound Ointment (MEBO)
- Standard of Care (Active Comparator): Topical application twice a day
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: MEBO Wound Ointment (MEBO) — Topical application twice a day
  Other Names: MEBO
  Arms: MEBO Wound Ointment (MEBO)
Other: Standard of Care — Topical application twice a day
  Arms: Standard of Care

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of MEBO in the treatment of subjects with diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
This is a phase II, randomized, controlled, multi-center study designed to assess the safety and efficacy of MEBO in the treatment of subjects with DFUs. Subjects meeting entry criteria will be randomly assigned in a 1:1 ratio for up to 8 weeks of treatment with either MEBO or SOC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Able and willing to provide informed consent
* Able and willing to comply with protocol visits and procedures
* Target ulcer duration of ≥4 weeks

Exclusion Criteria:

* Ulcer of a non-diabetic pathophysiology
* Known or suspected allergies to any of the components of MEBO
* Malignancy on target ulcer foot
* Non-compliance in the screening or run-in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The incidence of complete healing of the target ulcer. | 8 week treatment period

SECONDARY OUTCOMES:
Time required to achieve complete healing (days). | 8 week treatment period
Absolute and percentage change in ulcer surface area from baseline to endpoint. | 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Kirsner, MD, PhD, Study Chair — University of Miami
Locations (9):
- United States (9):
  - HOPE Research Institute, Phoenix, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - ILD Consulting, Inc., Encinitas, California
  - Sacramento Foot and Ankle Center, Fair Oaks, California
  - Valley Vascular Surgery Associates, Fresno, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Complete Family Foot Care, McAllen, Texas
  - Endeavor Clinical Trials, San Antonio Podiatry Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No